CLINICAL TRIAL: NCT04184271
Title: Pharmacokinetics of Advantage Arrest
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Advantage Silver Dental Arrest, LLC (Industry)
Collaborators: University of Washington (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016-11-08
Record Dates: First submitted 2019-11-28; First posted 2019-12-03 (Actual); Results first posted 2020-08-14 (Actual); Last update posted 2021-01-26 (Actual); Status verified 2020-07

CONDITIONS: Dental Caries
Keywords: adult; fluoride; silver; silver diamine fluoride; pharmacokinetics
MeSH Terms: conditions — Dental Caries | interventions — silver diamine fluoride

STUDY DESIGN:
Intervention Model Description: Open label exposure--response study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 38% silver diamine fluoride (Experimental): 38% silver diamine fluoride, topical, 1 drop, single application
  Interventions: Drug: 38% silver diamine fluoride

INTERVENTIONS:
Drug: 38% silver diamine fluoride — Topical application of SDF to teeth
  Other Names: Advantage Arrest

SUMMARY:
The study aim is to characterize the kinetics of silver and fluoride after topical application of silver diamine fluoride.

DETAILED DESCRIPTION:
The purpose of this study is to characterize basic PK parameters (Cmax, t1/2, AUC, and total urinary recovery) to contribute to evidence for the safety of Advantage Arrest, consistent with Guidance for Industry--Exposure--Response Relationships (April 2003).

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older, minimum 20 teeth, healthy, not taking prescription or OTC medications

Exclusion Criteria:

* pregnant, weighed less than 50 kg, had oral mucositis or ulcerative lesions, known sensitivity to silver or fluoride

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2017-09-30 (Actual); Study Completion 2019-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Milgrom, DDS, Principal Investigator — University of Washington
Locations (1):
- University of Washington Institute of Translational Health Sciences, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lin YS, Rothen ML, Milgrom P. Pharmacokinetics of 38% topical silver diamine fluoride in healthy adult volunteers. J Am Dent Assoc. 2019 Mar;150(3):186-192. doi: 10.1016/j.adaj.2018.10.018. PMID 30803490

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 38% Silver Diamine Fluoride
Started | 16
Completed | 16
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | 38% Silver Diamine Fluoride
Number analyzed (Participants) | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.4 (13.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 15
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 11
  More than one race | 2
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 16
Silver Observed Baseline [Mean (Standard Deviation); unit: ng/mL] | 0.15 (0.03)
Baseline Fluoride [Mean (Standard Deviation); unit: ng/mL] | 26 (12)

OUTCOME MEASURES:

1. Primary Outcome: Observed Fluoride Urinary Recovery
Description: 24 hour fluoride urinary recovery (in mg)
Time Frame: baseline to 24 hours
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | 38% Silver Diamine Fluoride
Number analyzed (Participants) | 16
mg | 1.29 (0.81)

2. Primary Outcome: Observed Silver Tmax
Description: Observed silver time to maximum serum concentration in hours
Time Frame: baseline, 30 minutes, and 1, 2, 3, 4, 6, 8, 12, and 24 hours
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | 38% Silver Diamine Fluoride
Number analyzed (Participants) | 16
hours | 5.3 (5.8)

3. Primary Outcome: Observed Silver Cmax
Description: Observed silver maximum serum concentration in ng/mL
Time Frame: baseline, 30 minutes, and 1, 2, 3, 4, 6, 8, 12, and 24 hours
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | 38% Silver Diamine Fluoride
Number analyzed (Participants) | 16
ng/mL | 0.70 (0.52)

4. Primary Outcome: Observed Silver Baseline-Corrected Cmax
Description: Observed silver baseline-corrected maximum serum concentration in ng/mL
Time Frame: baseline, 30 minutes, and 1, 2, 3, 4, 6, 8, 12, and 24 hours
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | 38% Silver Diamine Fluoride
Number analyzed (Participants) | 16
ng/mL | 0.67 (0.49)

5. Primary Outcome: Observed Silver t1/2
Description: Observed silver serum elimination half-life in hours
Time Frame: baseline, 30 minutes, and 1, 2, 3, 4, 6, 8, 12, and 24 hours
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | 38% Silver Diamine Fluoride
Number analyzed (Participants) | 16
hours | 46 (26)

6. Primary Outcome: Observed Silver 24 Hour Urinary Concentration
Description: Observed silver 24-hour urinary concentration in ng/mL
Time Frame: baseline to 24 hours
Measure: Mean (Full Range); unit: ng/mL
Arm/Group | 38% Silver Diamine Fluoride
Number analyzed (Participants) | 16
ng/mL | 0.05 [0.05 to 0.06]

ADVERSE EVENTS:
Time Frame: 24 hours
Arm/Group | 38% Silver Diamine Fluoride
All-Cause Mortality (participants affected / at risk) | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16
Other Adverse Events (participants affected / at risk) | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Statistical Analysis Plan (2020-07-30): https://cdn.clinicaltrials.gov/large-docs/71/NCT04184271/SAP_001.pdf
  • Study Protocol (2016-11-08): https://cdn.clinicaltrials.gov/large-docs/71/NCT04184271/Prot_002.pdf